CLINICAL TRIAL: NCT04923542
Title: Phase I/II Study of Stereotactic Radiation and Abemaciclib in the Management of Hormone Receptor Positive HER2 Negative Breast Cancer Brain Metastases
Brief Title: Stereotactic Radiation & Abemaciclib in the Management of HR+/HER2- Breast Cancer Brain Metastases
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MCC-20899
Record Dates: First submitted 2021-06-08; First posted 2021-06-11 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Brain Metastases; HR+ Metastatic Breast Cancer
MeSH Terms: conditions — Brain Neoplasms | interventions — Radiosurgery; abemaciclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase 1: Radiation Therapy and Abemaciclib (Experimental): Treatment will be initiated with one week of abemaciclib followed by stereotactic radiation to sites of brain metastases or post-operative cavities with continued abemaciclib. In the phase I portion, safety will be monitored initially by a 3+3 design. If unexpected neurologic toxicities are noted, the dose of radiation therapy will be modified.
  Interventions: Radiation: Stereotactic Radiosurgery (SRS); Drug: Abemaciclib; Drug: Endocrine therapy
- Phase 2: Radiation Therapy and Abemaciclib (Experimental): Treatment will be initiated with one week of abemaciclib followed by stereotactic radiation at the phase 1 dose to sites of brain metastases or post-operative cavities with continued abemaciclib.
  Interventions: Radiation: Stereotactic Radiosurgery (SRS); Drug: Abemaciclib; Drug: Endocrine therapy

INTERVENTIONS:
Radiation: Stereotactic Radiosurgery (SRS) — Patients will receive single session SRS to intact brain metastases and post-operative cavities. For intact brain metastases, this will be 15 Gy to lesions between 31-40 mm, 18 Gy to 21- 30 mm, and 24 Gy to lesions measuring ≤ 20 mm.
Drug: Abemaciclib — Abemaciclib is an orally administered selective small-molecule inhibitor of CDK4 and CDK6 that is 14 times more potent against CDK4 than CDK6 in enzymatic assays that is approved for the treatment of advanced or metastatic breast cancers. Abemaciclib will be administered at a dose of 150 mg twice daily.
  Other Names: Verzenio; Ramiven
Drug: Endocrine therapy — Abemaciclib will be administered with standard of care endocrine therapy. Endocrine therapy can consist of fulvestrant or an aromatase inhibitor. Dosing of concurrent endocrine therapy with abemaciclib should follow standard dosing and safety guidelines.
  Other Names: hormone therapy

SUMMARY:
This is a single arm study of abemaciclib and endocrine therapy with stereotactic radiosurgery (SRS) among patients with hormone receptor (HR)+/HER2- metastatic breast cancer brain metastases.

DETAILED DESCRIPTION:
The study is designed as a prospective, single-arm, nonrandomized, open-label, phase I/II trial of abemaciclib and endocrine therapy with stereotactic radiosurgery (SRS) among patients with hormone receptor (HR)+/HER2- metastatic breast cancer brain metastases. Treatment will be initiated with one week of abemaciclib followed by stereotactic radiation to sites of brain metastases or post-operative cavities with continued abemaciclib. Safety will be monitored initially by a 3+3 design. This will be followed by a phase 2 study to evaluate intracranial progression free survival (PFS). If unexpected neurologic toxicities are noted, the dose of radiation therapy will be modified.

ELIGIBILITY:
Inclusion Criteria:

* HR+ breast cancer to fulfill the requirement of HR+ disease, a breast cancer must express (≥ 1%), by immunohistochemistry (IHC), at least 1 of the hormone receptors (estrogen receptor [ER] or progesterone receptor [PR]) as defined in the American Society of Clinical Oncology (ASCO) / College of American Pathologists (CAP) Guidelines
* To fulfill the requirement of HER2- disease, a breast cancer must not demonstrate, at initial diagnosis or upon subsequent biopsy, overexpression of HER2 by either IHC or in-situ hybridization as defined by the ASCO / CAP Guidelines
* ≤ 15 brain metastases eligible for stereotactic radiation
* Able to swallow oral medications
* Willing to comply with all study procedures and available for duration of the study
* Measurable brain disease per RANO-BM criteria that can be measured in at least one dimension as ≥ 0.5 cm for both intact brain metastases and post-operative cavities
* Eligible for SRS to brain metastases or to the post-operative bed following surgical resection
* Maximum diameter of the largest intact brain metastases ≤ 4 cm
* Eastern Cooperative Oncology Group performance status 0 to 2
* A formalin-fixed, paraffin-embedded tumor tissue block or 10 unstained slides of intracranial/extracranial tumor sample (archival or recent) for biomarker evaluation should be made available and submitted to the central lab for correlative studies. If attempts to obtain archival tissue are unsuccessful the patient may be enrolled.
* Individuals with prior SRS/fractioned stereotactic radiotherapy (FSRT) treatment will be allowed if active measurable disease has not previously been treated with radiation therapy
* Women of childbearing potential (WOCBP) must have a negative serum pregnancy test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin) within 7 days of the first dose of abemaciclib
* WOCBP must agree to follow instructions for method(s) of contraception for the duration of treatment with study drug(s), and for three weeks following the last dose of abemaciclib
* Adequate organ function as defined in protocol

Exclusion Criteria:

* Presence of leptomeningeal disease
* Prior receipt of whole brain radiation therapy
* Prior receipt of abemaciclib in the setting of brain metastases or in the past 6 months for the treatment of metastatic disease.
* All toxicities attributed to prior anticancer therapy must have been resolved to Grade 1 (NCI CTCAE Version 5) or baseline before administration of study drug(s) other than: a. Toxicities attributed to prior anticancer therapy that either are not expected to resolve and/or result in long-lasting sequelae, such as neuropathy after platinum-based therapy b. Toxicities that are not expected to interfere with study treatment, such as fatigue, alopecia, or grade 2 hematologic toxicity
* Women who are pregnant or breastfeeding
* The patient has serious and/or uncontrolled preexisting medical condition(s) that, in the judgment of the investigator, would preclude participation in this study (for example, interstitial lung disease, severe dyspnea at rest or requiring oxygen therapy, severe renal impairment [e.g. estimated creatinine clearance <30ml/min], history of major surgical resection involving the stomach or small bowel, or preexisting Crohn's disease or ulcerative colitis or a preexisting chronic condition resulting in baseline Grade 2 or higher diarrhea)
* The patient has active systemic bacterial infection (requiring intravenous [IV] antibiotics at time of initiating study treatment), fungal infection, or detectable viral infection (such as known human immunodeficiency virus positivity or with known active hepatitis B or C [for example, hepatitis B surface antigen positive]. Screening is not required for enrollment
* The patient has a personal history of any of the following conditions: syncope of cardiovascular etiology, ventricular arrhythmia of pathological origin (including, but not limited to, ventricular tachycardia and ventricular fibrillation), or sudden cardiac arrest
* History of prior malignancy within 2 years prior to screening, with the exception of those with a negligible risk of metastasis or death (e.g., 5-year OS of >90%), such as but not limited to, non-melanoma skin carcinoma, or stage I endometriod uterine cancer, and others at the discretion of the PI.
* Major surgery or significant traumatic injury that has not been recovered from by 14 days before the initiation of study drug
* Current or prior participation in a study of an investigational agent or investigational device within 2 weeks of first dose of study treatment
* History of allergy or hypersensitivity to any of the study drugs or study drug components
* Prisoners or individuals who are involuntarily incarcerated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Estimated)
Dates: Start 2021-11-30 (Actual); Primary Completion 2026-11-05 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Intracranial Progression Free Survival (PFS) | Up to 12 months
  Intracranial Progression Free Survival: defined as the time from the date of start of treatment to investigator-determined date of progression or death due to any cause, whichever comes first. Progression will be determined by Response Assessment in Neuro-Oncology Brain Metastases (RANO-BM) Criteria.

SECONDARY OUTCOMES:
Intracranial local brain tumor control | Up to 12 months
  Intracranial local brain tumor control following SRS and abemaciclib will be determined from irradiated lesions according to RANO-BM criteria.
Intracranial distant brain tumor control | Up to 12 months
  Intracranial distant brain tumor control following SRS and abemaciclib will determined by the development of new lesions outside of the irradiated area.
Extracranial Progression Free Survival | Up to 12 months
  Extracranial Progression Free Survival: Time from the date of start of treatment to the investigator determined date of progression (determined by RECIST) or death due to any cause, whichever occurs first.
Overall Survival | Up to 12 months
  Overall Survival is defined as the time from the start of treatment to death due to any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Kamran A Ahmed, MD, Principal Investigator — Moffitt Cancer Center; Heather Han, MD, Principal Investigator — Moffitt Cancer Center
Locations (2):
- United States (2):
  - Moffitt Cancer Center, Tampa, Florida
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Moffitt Cancer Center's Clinical Trials Website — https://moffitt.org/clinical-trials-research/clinical-trials/?source=footer